CLINICAL TRIAL: NCT02796625
Title: Development of a Reliable Neurophysiological Pain Assessment Tool: Alpha as a Predictive Biomarker
Brief Title: Alpha as a Predictive Biomarker
Acronym: APB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Purdue Pharma LP (Industry)
Responsible Party: Principal Investigator, David Seminowicz, Associate Professor, Department of Neural and Pain Sciences, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10017571
Record Dates: First submitted 2016-05-25; First posted 2016-06-13 (Estimated); Results first posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-07

CONDITIONS: Pain
Keywords: EEG; healthy subjects
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Painful Stimuli (Experimental): Participants will be exposed to painful heat
  Interventions: Other: Painful Stimuli

INTERVENTIONS:
Other: Painful Stimuli — warm or painful heat administration

SUMMARY:
The investigators will use non-invasive recordings of brain activity to measure pain as a proxy to self-report. Participants will undergo testing for about 3 hours on two separate days. The testing will involve experiencing painful heat.

DETAILED DESCRIPTION:
Neurophysiological investigations of pain have suggested that electroencephalograph (EEG) measures of peak alpha frequency might provide a means of pain assessment. In healthy subjects, increased peak alpha frequency is strongly correlated with pain self-reports after exposure to acute noxious heat. Conversely, chronic pain patients compared to healthy control display decreased peak alpha frequencies higher in alpha power. Measures of peak alpha frequency also show a negative relationship with disease duration, suggesting that peak alpha frequency may not only index ongoing pain but also disease progression. The overall aim is to determine the predictive accuracy, reliability, and specificity of EEG alpha activity in acute pain and a model of neuropathic pain in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak, read, and write English
* Between 21 and 44 years of age
* Able to understand and willing to comply with all study procedures and is available for the duration of the study
* Free of an acute or chronic pain condition
* Not history of psychiatric or neurologic condition

Exclusion Criteria:

* Unable to undergo EEG, assessed on an individual basis
* History of unstable major psychiatric disorder (self-report)
* History of chronic pain (self-report)
* More than 14 alcoholic drinks per week on average (self-report)
* Active [within 6 months] substance or alcohol abuse (self-report and urine toxicology)
* Use of opioids (self-report and urine toxicology)
* History of major depressive disorder (self-report)
* Pregnant or Lactating (women only), based on (self-report and urine test)
* Anything that, in the opinion of the investigator, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study
* Uncontrolled (systolic blood pressure > 175 mmHg or diastolic blood pressure >105 mmHg) or unstable hypertension

Ages: 21 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Seminowicz, PhD, Principal Investigator — University of Maryland Dental School
Locations (1):
- University of Maryland School of Dentistry, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Painful Stimuli
Started | 80
Completed | 61
Not Completed | 19

BASELINE CHARACTERISTICS:
Arm/Group | Painful Stimuli
Number analyzed (Participants) | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 61
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 27.8 [21 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 61

OUTCOME MEASURES:

1. Primary Outcome: Peak Alpha Frequency (Hz)
Description: The highest power of EEG-based alpha activity in the 8-12Hz frequency range, calculated using the center of gravity method.
Time Frame: pain-free and pain states at the baseline visit
Population: all participants with valid data
Measure: Mean (Standard Deviation); unit: frequency (Hz)
Arm/Group | Painful Stimuli
Number analyzed (Participants) | 61
frequency (Hz) | 10.04 (0.20)

2. Secondary Outcome: Alpha Wave Activity Reliability
Time Frame: alpha activity at pain-free and pain states, assessed at a second visit following the first visit by at least 3 week
Population: Participants with data at visits 1 and 2
Measure: Number; unit: Spearman rho
Arm/Group | Painful Stimuli
Number analyzed (Participants) | 43
Spearman rho | .81

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Painful Stimuli
All-Cause Mortality (participants affected / at risk) | 0/61
Serious Adverse Events (participants affected / at risk) | 0/61
Other Adverse Events (participants affected / at risk) | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT02796625/Prot_SAP_000.pdf